CLINICAL TRIAL: NCT03179397
Title: A Clinical Trial to Evaluate the Safety and Effectiveness of Model SC9 Silicone IOL for the Visual Correction of Aphakia Secondary to the Removal of a Cataractous Lens in Adult Patients With or Without Presbyopia
Brief Title: Clinical Trial to Evaluate the Model SC9 IOL Compared to the Model LI61SE IOL (Bausch & Lomb)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor did not recruit enough subjects to file PMA.
Sponsor: CORD, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SC9-0015
Record Dates: First submitted 2017-05-29; First posted 2017-06-07 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Masking Description: Enrolled subjects will not be told which IOL they have received until the end of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Model SC9 (Experimental): Investigational IOL
  Interventions: Device: Model SC9
- Model LI61SE (Active Comparator): FDA Approved IOL
  Interventions: Device: Model LI61SE

INTERVENTIONS:
Device: Model SC9 — Experimental
  Arms: Model SC9
Device: Model LI61SE — Active Comparator
  Arms: Model LI61SE

SUMMARY:
To evaluate the Model SC9 Intraocular Lens for the improvement of near and intermediate vision when compared to a legally marketed monofocal IOL.

DETAILED DESCRIPTION:
Subjects will be randomized to one of two groups. Group A, (Test Lens, Model SC9) or Group B, (Control Lens, Model LI61SE, Bausch and Lomb).

Both groups will be randomized to receive either unilateral or bilateral implantation. No bilateral implantation is allowed in Phase 1. (50 subjects).

Subjects will be followed for 36 Months.

ELIGIBILITY:
Inclusion Criteria:

* Twenty-two years or older at the time of surgery and diagnosed with bilateral cataracts
* Able to comprehend and sign a statement of informed consent
* Willing and able to complete all required postoperative visits
* Calculated Lens Power within the available range for the study IOL's
* Planned cataract removal by phacoemulsification
* Potential postoperative visual acuity of BCDVA 0.2 LogMAR (20/32) or better in both eyes
* Subjects with less than 1.0D of corneal astigmatism
* Clear intraocular media other than cataract in the study eye
* Preoperative BCDVA worse than 0.2 LogMar (20/32) with or without glare
* Pupil size greater or equal to 6.0mm after dilation

Exclusion Criteria:

* Any corneal abnormality, other than regular corneal astigmatism
* Subjects with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal disorders) that are predicted to cause future acuity losses to a level worse than 0.2 LogMAR (20/32)
* Previous refractive surgery
* Amblyopia
* Clinical severe corneal dystrophy (e.g., epithelial, stromal, or endothelial dystrophy)
* Diabetic retinopathy
* Extremely shallow anterior chamber, not due to swollen cataract
* Microphthalmos
* Previous retinal detachment
* Previous corneal surgery
* Recurrent severe anterior or posterior segment inflammation of unknown etiology
* Rubella or traumatic cataract
* Iris Neovascularization
* Glaucoma (uncontrolled or controlled with medication)
* Aniridia
* Optic nerve atrophy
* Damaged incomplete zonules
* Systemic disease that could increase the operative risk or confound the outcome
* Medications that, in the opinion of the investigator may confound the outcome or increase the risk to the subject (tamsulosin hydrochloride (Flomax) or other medications with similar side-effects (floppy iris syndrome)

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Improvement in Visual Acuity Measurements using the LogMar Scale | 12 Months
  Subjects must read 20/40 or better, distance corrected near visual acuity and 20/40 or better distance corrected intermediate visual acuity. This is achieved with the subject wearing their best corrected spectacle correction in place and reading a series of letters at 40cm/16" and 80cm/32". Total letters read for each line will determine their visual acuity

SECONDARY OUTCOMES:
Defocus testing in 0.5D increments from -0.5 to -5.00D | 12 Months
  A sub-set of 50 subjects will undergo defocus testing with their best distance correction in place. Minus Lenses in 0.5D increments will be placed over their best spectacle correction. Total letters read for each diopter will be recorded. Percentage of eyes with improvement of monocular depth of focus by at least 0.5D mean difference between the Model SC9 and control lens.(significance level of 0.025). To demonstrate superiority of at least 0.5D compared to the control lens >75% of eyes implanted with the Model SC9 should demonstrate superiority by at least 0.5D mean difference compared to the control lens.

CONTACTS AND LOCATIONS:
Overall Officials: John Hovanesian, M.D., Study Chair — CORD, LLC
Locations (13):
- United States (13):
  - Davies Eye Center, Carlsbad, California
  - Harvard Eye Associates, Laguna Hills, California
  - Coastal Vision Laser Eye Center, Orange, California
  - Shasta Eye Medical Group, Inc., Redding, California
  - Aker-Kasten Eye Center, Boca Raton, Florida
  - The Eye Institute of West Florida, Largo, Florida
  - Chu Vision Institute, Bloomington, Minnesota
  - Silverstein Eye Centers, Kansas City, Missouri
  - Center for Sight, Las Vegas, Nevada
  - Fine, Hoffman and Sims, Eugene, Oregon
  - Houston Eye Associates, Houston, Texas
  - Parkhurst NuVision, San Antonio, Texas
  - Eye Associates of South Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No